CLINICAL TRIAL: NCT04439214
Title: MATCH Treatment Subprotocol Z1D: Nivolumab in Patients With Tumors With Mismatch Repair Deficiency
Brief Title: Testing Nivolumab as a Potential Targeted Treatment in Cancers With Mismatch Repair Deficiency (MATCH-Subprotocol Z1D)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-03172; NCI-2020-03172 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-Z1D (Other: ECOG-ACRIN Cancer Research Group); EAY131-Z1D (Other: CTEP); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Results first posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Plasma Cell Myeloma
Keywords: Nivolumab; Lymphoma; Mismatch repair deficiency
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Multiple Myeloma; Turcot syndrome | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (nivolumab) (Experimental): Patients receive nivolumab IV over 30-60 minutes on days 1 and 15 of cycles 1-4 and on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase II MATCH treatment trial identifies the effects of nivolumab in patients whose cancer has a genetic change called mismatch repair deficiency. Mismatch repair deficiency refers to cells that have mutations (changes) in certain genes that are involved in correcting mistakes made when DNA is copied in a cell. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of cancer cells with mismatch repair deficiency to grow and spread. Researchers hope to learn if nivolumab will shrink this type of cancer or stop its growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression.

EXPLORATORY OBJECTIVES:

I. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

II. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive nivolumab intravenously (IV) over 30-60 minutes on days 1 and 15 of cycles 1-4 and on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months if less than 2 years from study entry, and then every 6 months for year 3 from study entry.

THE MATCH SCREENING TRIAL:

Please see NCT02465060 for information on the MATCH Screening Protocol and applicable documents.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol prior to registration to treatment subprotocol
* Patients must have mismatch repair deficiency as determined via the MATCH Master Protocol
* Women of childbearing potential (WOCBP) receiving nivolumab must agree to use adequate contraception (hormonal or double barrier method of birth control; abstinence) from one week prior to study treatment starting, during treatment, and for a period of 5 months after the last dose of nivolumab. Men receiving nivolumab and who are sexually active with WOCBP must agree to use adequate contraception (hormonal or double barrier method of birth control; abstinence) from one week prior to study treatment starting, during treatment, and for a period of 7 months after the last dose of nivolumab
* Patients with hepatitis B virus (HBV) or hepatitis C virus (HCV) infection may be eligible provided they have the following:

  * There must be no evidence of clinically significant hepatic injury from hepatitis virus infection
  * For HBV, patients must be on suppressive therapy and have undetectable HBV viral load
  * For HCV, patients must either be on suppressive therapy for HCV or have already completed therapy thought to have eradicated HCV

Exclusion Criteria:

* Patients must not have known hypersensitivity to nivolumab or compounds of similar chemical or biologic composition
* No prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-OX-40, anti-CD40 or anti-CTLA-4 antibodies (or any other antibody targeting T cell co-regulatory pathways)
* Patients with cancers for which nivolumab is approved or becomes approved are excluded (e.g: colorectal cancer, locally advanced or metastatic urothelial carcinoma, unresectable or metastatic melanoma, metastatic non-small cell lung cancer, advanced renal cell carcinoma, classical Hodgkin lymphoma, and recurrent or metastatic squamous cancer of the head and neck)
* Must not have received any of the following therapies within four weeks prior to the first dose of the study drug: IL-2, interferon, or other non-study immunotherapy regimens or immunosuppressive agents
* Must not have a history of toxic epidermal necrolysis (Stevens-Johnson syndrome)
* Must not have received growth factors, including but not limited to granulocyte-colony stimulating factor (G-CSF), granulocyte macrophage-colony stimulating factor (GM-CSF), erythropoietin, etc. within 2 weeks of study drug administration. Use of such agents while on study is also prohibited. Prior use of growth factors should be documented in the patient's medical history
* Must not have a history of any autoimmune disease: inflammatory bowel disease, (including ulcerative colitis and Crohn's disease), rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus (SLE) autoimmune vasculitis (e.g., Wegener's Granulomatosis), central nervous system (CNS) or motor neuropathy considered to be of autoimmune origin (e.g., Guillain-Barre syndrome, myasthenia gravis, multiple sclerosis). Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event). Entry of patients with autoimmune diagnoses not listed here must be approved by the protocol chair
* Must not be on supplemental home oxygen
* Must not have evidence of interstitial lung disease
* Patients with a requirement for steroid treatment or other immunosuppressive treatment: Patients will be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* No history of severe hypersensitivity reaction to any monoclonal antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2020-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nilofer S Azad, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Azad NS, Gray RJ, Overman MJ, Schoenfeld JD, Mitchell EP, Zwiebel JA, Sharon E, Streicher H, Li S, McShane LM, Rubinstein L, Patton DR, Williams PM, Coffey B, Hamilton SR, Bahary N, Suga JM, Hatoum H, Abrams JS, Conley BA, Arteaga CL, Harris L, O'Dwyer PJ, Chen AP, Flaherty KT. Nivolumab Is Effective in Mismatch Repair-Deficient Noncolorectal Cancers: Results From Arm Z1D-A Subprotocol of the NCI-MATCH (EAY131) Study. J Clin Oncol. 2020 Jan 20;38(3):214-222. doi: 10.1200/JCO.19.00818. Epub 2019 Nov 25. PMID 31765263

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subprotocol Z1D was activated in NCI-MATCH on May 31, 2016. Patients enrolled for screening by the MATCH assay between this date and the end of screening enrollment in May 2017, were evaluated for MSH2 and MLH1 expression by immunohistochemistry (IHC). In the end, 47 patients were enrolled to the subprotocol.
Pre-assignment Details: To be assigned to a specific MATCH subprotocol, patients needed to submit a tumor biopsy for molecular characterization and those with molecular variants addressed by treatments included in the trial entered corresponding MATCH subprotocol. For the subprotocol Z1D, patients had to have complete loss of nuclear expression of MLH1 or MSH2 MMR gene products by IHC.
Period: Overall Study
Arm/Group | Treatment (Nivolumab)
Started | 47
Eligible | 42
Treated | 47
Treated and Reported Adverse Event Data | 46 (One patient experienced disease progression in cycle 1 and an AE form was not submitted.)
Eligible and Treated | 42
Completed (Treatment continued until progression or intolerability. At the time of the final analysis of the data, 9 patients were still receiving protocol treatment.) | 0
Not Completed | 47
Not completed — Adverse Event | 13
Not completed — Disease progression | 16
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2
Not completed — Declining health | 1
Not completed — Still receiving treatment at the time of the analysis | 9
Not completed — Ineligible | 5

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 42
Age, Continuous [Median (Full Range); unit: years] | 60.5 [44 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 35
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate was defined as the proportion of patients with best overall response of complete response (CR) or partial response (PR) among all eligible and treated patients. Best overall response was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. The 90% two-sided binomial exact confidence interval was calculated for ORR.
Time Frame: assessed at baseline, then every 8 weeks for the first 2 years, then every 12 weeks in year 3, until disease progression
Population: Eligible and treated patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 42
percentage of participants | 35.7 [23.5 to 49.5]

2. Secondary Outcome: 6-month Progression-free Survival (PFS) Rate
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. The 6-month PFS rate was estimated using the Kaplan-Meier method which can provide a point estimate for any specific time point. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients.
Time Frame: as for outcome 1
Population: Eligible and treated patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 42
percentage of participants | 51.3 [38.2 to 64.5]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients.
Time Frame: as for outcome 1
Population: Eligible and treated patients
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 42
months | 6.3 [3.4 to 13.3]

ADVERSE EVENTS:
Time Frame: Assessed every 28 days while on treatment and for 30 days after the end of treatment, up to 3 years
Description: All the 47 enrolled patients started protocol therapy and followed for survival, but 1 patient had disease progression in cycle 1 and adverse event data were not reported. So adverse events were reported for the 46 patients who reported adverse event data, and all-cause mortality was reported for the 47 patients.
Arm/Group | Treatment (Nivolumab)
All-Cause Mortality (participants affected / at risk) | 24/47
Serious Adverse Events (participants affected / at risk) | 20/46
Other Adverse Events (participants affected / at risk) | 40/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Nivolumab) (N=46)
Anemia (Blood and lymphatic system disorders) | 8
Fatigue (General disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Creatinine increased (Investigations) | 2
Ejection fraction decreased (Investigations) | 1
Weight gain (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Myelitis (Nervous system disorders) | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1
Hypotension (Vascular disorders) | 1
Peripheral ischemia (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Nivolumab) (N=46)
Anemia (Blood and lymphatic system disorders) | 12
Edema limbs (General disorders) | 3
Fatigue (General disorders) | 21
Pruritus (Skin and subcutaneous tissue disorders) | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8
Hyperthyroidism (Endocrine disorders) | 7
Hypothyroidism (Endocrine disorders) | 7
Diarrhea (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 6
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 6
Creatinine increased (Investigations) | 3
Lymphocyte count decreased (Investigations) | 6
Platelet count decreased (Investigations) | 6
White blood cell decreased (Investigations) | 3
Investigations - Other, specify (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 7
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 4
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Hot flashes (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT04439214/Prot_001.pdf